CLINICAL TRIAL: NCT06946420
Title: SENECA: First Line metaStatic pancrEatic caNcer Primary and Distant (if Oligometastatic) lEsion direCted rAdiotherapy, a Phase III Randomized Multicentric Trial
Brief Title: SENECA: First Line metaStatic pancrEatic caNcer Primary and Distant (if Oligometastatic) lEsion direCted rAdiotherapy
Acronym: SENECA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Manfrida Stefania, Medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001898 24
Record Dates: First submitted 2025-03-26; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Radiation Therapy; SBRT; Pancreatic Cancer Metastatic
MeSH Terms: interventions — Radiosurgery; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard systemic therapy (chemotherapy) without RT/SBRT (Other): Patients will undergo only standard systemic treatment (chemotherapy drugs at the discretion of the oncologist) without receiving radiotherapy or stereotactic treatment.
  Interventions: Drug: Standard systemic therapy (chemotherapy) without RT/SBRT
- RT / SBRT before standard systemic therapy (chemotherapy) (Experimental): Combination of RT on primary pancreatic Gross Tumor Volume (GTV) (SBRT or RT) + SBRT on each of the distal lesions SBRT or RT will be delivered immediately before the initiation of systemic therapy ((chemotherapy drugs at the discretion of the oncologist))
  Interventions: Radiation: SBRT or RT on primary pancreatic and/or metastatic distant lesions before chemotherapy

INTERVENTIONS:
Radiation: SBRT or RT on primary pancreatic and/or metastatic distant lesions before chemotherapy — This group of patients will first undergo radiotherapy on the primary pancreatic lesion and stereotactic treatment on the metastatic sites before being started on standard systemic therapy (chemotherapy)
  Other Names: SBRT; Radiation therapy; pancreatic cancer
  Arms: RT / SBRT before standard systemic therapy (chemotherapy)
Drug: Standard systemic therapy (chemotherapy) without RT/SBRT — This group of patients will undergo standard systemic therapy (chemotherapy drugs chosen by oncologist) without radiotherapy treatment
  Other Names: systemic therapy; No radiation; standard
  Arms: Standard systemic therapy (chemotherapy) without RT/SBRT

SUMMARY:
Thisi is an Interventional drug-free randomized 1:1 open-label, multicenter, phase 3 trial in patients with first-line metastatic pancreatic cancer. The interventional group of patients will undergo radiotherapy on the primary lesion and SBRT on distal metastatic sites before receiving standard systemic therapy (chemotherapy), while the other group of patients will receive only standard systemic therapy (chemotherapy) without undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer, metastatic, candidate for first-line treatment standard systemic; either newly diagnosed in metastatic stage or first progression to metastasis.
* Obtaining informed consent
* Patients >18 years of age
* ECOG 0-2
* Performance of imaging (CT with mdc, MRI with mdc, CT-PET with appropriate tracer) adequate for baseline local and systemic staging and likely to be similarly repeatable at 6 and 12 months after randomization
* Confirmation at the time of randomization, by the Radiotherapy Center, that it is possible to perform all treatments potentially planned for the patient (if enrolled in experimental arm) within a maximum of 25 total days prior to referral to the Medical Oncology Center for systemic therapy

Exclusion Criteria:

* Metastatic picture of line subsequent to the first
* Technical or organizational impracticality to the eventual termination of radiation treatments Within 25 days after randomization
* Inability to express independent consent to treatments
* Pregnancy
* Patient in hospice or with prognosis < 6 months
* Predicted unavailability for follow-up at 6 months
* Absence of adequate or likely non-repeatable pretreatment imaging study at 6 and 12 months
* Previous radiation therapy
* Previous radiometabolic therapy
* Inability to maintain treatment position for SBRT
* Symptomatic emergent or other presentation precluding study development as planned (e.g., epidural compression of the spinal cord or cauda equina)
* Previous chemotherapy, immunotherapy or target therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2030-01-10 (Estimated); Study Completion 2031-01-10 (Estimated)

PRIMARY OUTCOMES:
Absence of symtomps | From the week after the treatment up to 12 months after
  Comparison between the experimental arm and the standard arm in terms of pain reduction or absence of pain (particularly with regard to abdominal pain and widespread pain from disease) using NRS scale, one-dimensional 11-point scale that assesses pain intensity in adult

SECONDARY OUTCOMES:
Pain level | From the week after the treatment up to 12 months after
  Level of metastasis-associated or primary pain (presence/absence, level and response)
Radiotherapy use | From the week after the treatment up to 12 months after
  Rate of recourse to Radiotherapy for pain, obstruction, bleeding or other symptom referable to the primary at 6 months from randomization (and not present at randomization)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Agostino Gemelli IRCSS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided